CLINICAL TRIAL: NCT00398515
Title: A Phase I Trial of CC-5013 (Lenalidomide) and CCI-779 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Lenalidomide and Temsirolimus in Treating Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00151; NCI-2009-00151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-2006C0040; CDR0000514831; OSU-05115; 05115 (Other: Ohio State University Medical Center); 7314 (Other: CTEP); U01CA076576 (NIH); NCT01645553 (obsolete NCT alias); NCT01664442 (obsolete NCT alias)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Refractory Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; temsirolimus; Sirolimus

ARMS (1):
- Treatment (antiangiogenesis, chemotherapy, enzyme inhibitor) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22 and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Drug: temsirolimus; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus when given together with lenalidomide in treating patients with previously treated multiple myeloma. Lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Drugs used in chemotherapy, such as temsirolimus, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Temsirolimus may also stop the growth of cancer cells by blocking some of the enzymes needed for their growth. Giving lenalidomide together with temsirolimus may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of CCI-779 (temsirolimus) when given together with lenalidomide in patients with previously treated multiple myeloma.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. II. Determine the clinical response of patients treated with this regimen. III. Determine the pharmacokinetics of this regimen. IV. Determine the pharmacodynamic effects of this regimen in these patients. V. Determine the effect of this regimen on immunological cellular and serological parameters and hematopoietic precursor cells.

OUTLINE: This is a dose-escalation study of CCI-779.

Patients receive temsirolimus intravenously (IV) over 30 minutes on days 1, 8, 15, and 22 and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving at least a partial response after 12 courses may continue to receive CCI-779 and lenalidomide as above in the absence of disease progression. Cohorts of 3 patients receive escalating doses of CCI-779 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Ten patients are treated at the MTD. Patients undergo blood sample and bone marrow collection periodically during study treatment for pharmacokinetic and pharmacodynamic studies, and to determine the immunomodulatory effects of CCI-779 and lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (MM)

  * Salmon-Durie stage IIA or IIIA
  * No stage B disease
* Meets ≥ 1 major AND 1 minor criterion OR ≥ 3 minor criteria

  * The following are considered major criteria:

    * Plasmacytoma on tissue biopsy
    * Bone marrow plasmacytosis with ≥ 30% plasma cells
    * Monoclonal paraprotein ≥ 3,500 mg/dL (IgG) or ≥ 2,000 mg/dL (IgA) OR monoclonal protein (Bence-Jones protein) ≥ 1,000 mg by 24-hour urine collection
  * The following are considered minor criteria:

    * Bone marrow plasmacytosis 10-29% of marrow cellularity
    * Monoclonal globulin spike < 3,500 mg/dL (IgG) or < 2,000 mg/dL (IgA)
    * Lytic bone lesions
    * Decrease in normal IgM (< 50 mg/dL), IgA (< 100 mg/dL), or IgG (< 600 mg/dL)
* Disease progression after ≥ 1 prior systemic treatment regimen* for MM (e.g., chemotherapy, high-dose corticosteroids, thalidomide, or bortezomib), defined as > 25% increase in serum or urine M-protein
* No solitary plasmacytoma
* No non-secretory MM (absent serum or urinary M-protein)
* ECOG performance status 0-2
* Life expectancy > 6 months
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Creatinine ≤ 2.0 mg/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Fasting cholesterol ≤ 350 mg/dL
* Fasting triglycerides ≤ 400 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception
* Must agree not to donate blood, sperm, or ova during and for 4 weeks after completion of study treatment
* No other prior or concurrent malignancy or myelodysplasia except for the following:

  * Basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Localized cancer treated with surgery only with no evidence of disease for > 5 years
* No history of recurrent deep vein thrombosis (DVT)/pulmonary embolism (PE) or DVT/PE occurring while on therapeutic levels of anticoagulation

  * Patients with DVT/PE within the past 6 months are eligible provided they receive full anticoagulation during study treatment
* No active infection requiring oral or intravenous antibiotics
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study compliance
* No known hepatitis B or C
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to lenalidomide or CCI-779
* See Disease Characteristics
* Prior lenalidomide allowed
* Prior high-dose chemotherapy with stem cell transplantation allowed
* More than 4 weeks since prior chemotherapy or other antimyeloma systemic therapy (e.g., thalidomide, bortezomib, or high-dose corticosteroids) and recovered
* No prior exposure to both lenalidomide and mTOR inhibitors (given together)

  * Treatment with single-agent lenalidomide or single-agent mTOR inhibitor allowed
* No other concurrent investigational agents
* No concurrent corticosteroids unless for physiologic maintenance
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent myeloid growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-03; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of temsirolimus when given together with lenalidomide | Course 1 (first 28 days)
  The MTD is the dose level at which less than 2 out of 6 patients experience dose limiting toxicities (DLT). The National Cancer Institute Common Terminology Criteria for Adverse events (CTCAE) version 3.0 will used to characterize toxicities.

SECONDARY OUTCOMES:
Toxicity of lenalidomide and temsirolimus combination therapy in previously treated mulple myeloma patients | From the time of their first treatment with lenalidomide and temsirolimus
  Measured by NCI CTCAE version 3.0.
Pharmacokinetic analysis of lenalidomide | Baseline and days 1 and 22 (lenalidomide only) of course 1
  Plasma drug levels will be measured by liquid chromatography and tandem mass spectroscopy.
Pharmacodynamics of temsirolimus in peripheral blood mononuclear cells (PBMC) | Days 1 and 8 of course 1
  PBMC will be used to assess the phosphorylation status of p70S6K to evaluate the pharmacodynamic activity of each dose level. This will assist in determining the biologically active dose in the event that dose limiting toxicity is not observed. The analysis of p70^S6K and phospho (P)-p70^S6K will be assessed by Western blotting using specific antibodies. The expression level will be quantified by densitometry. The inhibition of P- p70S6K will be correlated with clinical endpoints and PK parameters.
Assessment of serum cytokines; IL-2, sIL-2R, TNF-alpha, IFN-gamma, IL-1 beta, IL-1Ra, GM-CSF, IL-8, IL-6, sIL-6R, MIP-1 alpha, VEGF, and b-FGF | Baseline and then every 4 weeks
  Assessed by ELISA.
Assessment of peripheral blood immune cell subsets | Baseline and then every 4 weeks
  We will investigate immune cell subsets by flow-cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States